CLINICAL TRIAL: NCT01455922
Title: A Phase 3, Randomized, Active Comparator, Double-Blind, Multi-Center Study to Compare the Efficacy, Safety and Tolerability of ITCA 650 to Glimepiride as Add-on Therapy to Metformin in Patients With Type 2 Diabetes
Brief Title: A Study to Evaluate ITCA 650 Compared to Glimepiride as Add on Therapy for the Treatment of Type 2 Diabetes
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITCA 650-CLP-112
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Last update posted 2012-12-25 (Estimated); Status verified 2012-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- ITCA 650 60 mcg/day (Experimental)
  Interventions: Drug: ITCA 650
- glimepiride (Active Comparator)
  Interventions: Drug: glimepiride

INTERVENTIONS:
Drug: ITCA 650 — ITCA 650 is exenatide in DUROS
  Arms: ITCA 650 60 mcg/day
Drug: glimepiride — glimepiride will be up-titrated to 8 mg/day over first 13 weeks
  Arms: glimepiride

SUMMARY:
Phase 3 study to examine treatment with ITCA 650 compared to glimepiride when added to metformin monotherapy in reducing HbA1c in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c between 7.5% - 10.5%
* on metformin monotherapy
* BMI between 25 & 45 kg/m2

Exclusion Criteria:

* On thiazolidinedione, sulfonylurea, DPP-4, alpha glucosidase inhibitor, meglitinides or insulin within last 3 months
* history of pancreatitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c | 52 weeks
  52-week Treatment Period followed by 52-week Extension Period

CONTACTS AND LOCATIONS:
Locations (1):
- Intarcia Therapeutics, Inc, Hayward, California, United States